CLINICAL TRIAL: NCT02817425
Title: A Efficacy and Tolerability Study of Uracil/Ftorafur/Leucovorin Combined With Oxaliplatin (TEGAFOX) Sequential S-1 or SOX Sequential S-1 and S-1 Monotherapy in the Treatment of Adjuvant Chemotherapy for Gastric Cancer
Brief Title: A Efficacy and Tolerability Study of TEGAFOX Sequential S-1 in the Treatment of Adjuvant Chemotherapy for Gastric Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Xiao Chen, MD, Head of department, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013078
Record Dates: First submitted 2015-06-08; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: S-1; Adjuvant Chemotherapy; TEGAFOX
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SOX Sequential S-1 Group (Active Comparator): Patients received chemotherapy with" oxaliplatin+ S-1 " for 6 months and sequential "S-1" for 6 months
  Interventions: Drug: SOX Sequential S-1
- SOX Group (Active Comparator): Patients received chemotherapy with" oxaliplatin+ S-1 " for 12 months
  Interventions: Drug: SOX
- TEGAFOX Sequential S-1 (Experimental): Patients received chemotherapy with" TEGAFOX (oxaliplatin+ Tegafur +Leucovorin Calcium) " for 6 months and sequential "S-1" for 6 months
  Interventions: Drug: TEGAFOX Sequential S-1.

INTERVENTIONS:
Drug: SOX Sequential S-1 — 8 cycles SOX followed by S-1 monotherapy until disease progression. S-1: 40 mg/m2 bid,po, day 1 ~14 (S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid) Oxaliplatin: 130 mg/m2 iv 2h,day 1.Every 21 days as a cycle.
  Arms: SOX Sequential S-1 Group
Drug: SOX — S-1: 40 mg/m2 bid,po, day 1 ~14 (S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid) Oxaliplatin: 130 mg/m2 iv 2h,day 1. Every 21 days as a cycle
  Arms: SOX Group
Drug: TEGAFOX Sequential S-1. — 6 cycles TEGAFOX followed by S-1 monotherapy until disease progression. S-1: 40 mg/m2 bid,po, day 1 ~14 (S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid) Oxaliplatin: 130 mg/m2 iv 2h,day 1. TF 1000 mg/m2 with calcium folinate 300 mg/m2 IV infusion from Day 1 to Day 5 Every 28 days as a cycle.
  Arms: TEGAFOX Sequential S-1

SUMMARY:
This study is designed to compare the three chemotherapy regimens(TEGAFOX Sequential S-1 or SOX Sequential S-1 or SOX non-Sequential S-1) for postoperative patients with gastric cancer, observe and record the efficacy and tolerance,to evaluate which regimen is better.

ELIGIBILITY:
Inclusion Criteria:

* 75≧Age≧18
* Histologically or cytologically confirmed gastrointestinal cancer
* Stage Ⅱ or Ⅲ or Ⅳ
* ECOG ≦2
* Accept the gastric cancer radical resection
* Life expectancy of at least three months
* Written informed consent to participate in the trial

Exclusion Criteria:

* History of severe hypersensitivity reactions to the ingredients of S-1\TF\5-FU/calcium folinate or oxaliplatin
* Inadequate hematopoietic function which is defined as below:

  * white blood cell (WBC) less than 5x10^9/L
  * absolute neutrophil count (ANC) less than 2x10^9/L
  * platelets less than 100*10^9/L
* Inadequate hepatic or renal function which is defined as below:

  * serum bilirubin greater than 2 times the upper limit of normal range
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULN if no demonstrable liver metastases or greater than 5 times the ULN in the presence of liver metastases
  * blood creatinine level greater than 2 times ULN
* Presence of peripheral neuropathy
* Receiving a concomitant treatment with other fluoropyrimidine drug or flucytosine drug
* Women who is pregnant or lactating or fertile women of child-bearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period (Including male)
* Psychiatric disorder or symptom that makes participation of the patient difficult;
* Concomitant illness that might be aggregated by active, non-controlled disease such as congestive heart failure, ischemic heart disease, uncontrolled hypertension or arrhythmia with in six months
* Severe complication(s), e.g., paresis of intestines, ileus, radiographically confirmed interstitial pneumonitis or pulmonary fibrosis, glomerulonephritis ,renal failure, poorly-controlled diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survial (OS) | Event driven, an expected average of 48 months

SECONDARY OUTCOMES:
Disease Free Survial | Event driven, an expected average of 24 months
Safety (Adverse Events) | Adverse events will be assessed at baseline (after the patients provided signed Informed Consent Form) until at least 4 weeks after the last dose of study drug was administered, an expected average of 3week
Dose intensity | Event driven, an expected average of 48 months
  Dose intensity will be used for present patients' compliance

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chen, MD, Principal Investigator — Second Hospital Affiliated to Lanzhou University
Locations (1):
- Second Hospital Affiliated to Lanzhou University, Lanzhou, Gansu, China